CLINICAL TRIAL: NCT02908282
Title: Topical Omega-3 Fatty Acids (REMOGEN® OMEGA) in the Treatment of Dry Eye
Acronym: REMOTOP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TRB Chemedica AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REMODES-DE-2015-12
Record Dates: First submitted 2016-09-13; First posted 2016-09-20 (Estimated); Last update posted 2018-08-15 (Actual); Status verified 2018-08

CONDITIONS: Dry Eye Syndromes
Keywords: tear film; omega-3 fatty acids; eye drops
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- PUFA (polyunsaturated fatty acids)-group (Other): REMOGEN OMEGA: Usage according to instructions for use.
  Interventions: Device: REMOGEN OMEGA
- C (control)-group (Other): Povidone: Usage according to instructions for use.
  Interventions: Device: Povidone

INTERVENTIONS:
Device: REMOGEN OMEGA — Lubricant eye drops: preservative-free, hypotonic microemulsion of polyunsaturated fatty acids and hydrating polymers provided in single-dose containers of 0.25 ml.
  Arms: PUFA (polyunsaturated fatty acids)-group
Device: Povidone — Artificial tears: preservative-free eye drops containing 2% povidone.
  Arms: C (control)-group

SUMMARY:
The primary objective of this study is to evaluate the efficacy of REMOGEN® OMEGA in reducing Dry Eye Syndrome (DES) symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patient between 18 and 80 years of age and in good general health condition.
* Signed written informed consent.
* Existence of moderate to severe DES symptoms defined as Break-up time (TBUT) ≤ 10 s (mean of 3 consecutive measurements) and OSDI questionnaire ≥ 20.

Exclusion Criteria:

* Contraindication for the use of the products (e.g. hypersensitivity to the constituents of the test products) or any study procedure.
* Concomitant or previous participation in a clinical investigation within the last 3 months.
* Concomitant therapies/manipulations that affect either the tear film, tear secretion or ocular surface integrity or would alter the effect of the devices being evaluated.
* Concurrent (systemic) DES-associated diseases that are not on a stable therapy since at least 1 month (therapy not expected to change)
* Glaucoma that is not on a stable dosage since at least 2 weeks (therapy not expected to change)
* Any diseases or characteristics judged by the investigator to be incompatible with the assessments and/or procedures for the study evaluation
* Pregnant or lactating females.
* Participants of childbearing age who do not use adequate methods of birth control.
* Subjects unable to understand the informed consent or having a high probability of noncompliance to the study procedures and/or non-completion of the study according to investigator's judgment (e.g. illiteracy, insufficient knowledge of local language).
* Subjects not capable of contracting and of understanding the nature, risks, significance and implications of the clinical investigation and unable to form a rational intention in the light of these facts.

Ages: 18 Years to 81 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2016-10; Primary Completion 2018-07 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
Ocular Surface Disease Index (OSDI©) questionnaire | Week 4
Tear film stability | Week 4
  Tear film breakup time (unit: seconds)

SECONDARY OUTCOMES:
OSDI questionnaire | Day 0, Week 12
Tear film stability | Day 0, Week 12
  Tear film breakup time (unit: seconds)
Visual acuity (best corrected) | Day 0, Week 4, Week 12
TearLab osmolarity test | Day 0, Week 4, Week 12
Inflammation marker matrix metalloproteinase 9 (MMP9) | Day 0, Week 4, Week 12
Lid-parallel conjunctival fold (LIPCOF) grading | Day 0, Week 4, Week 12
Corneal staining | Day 0, Week 4, Week 12
  Oxford grading scale
Tear volume | Day 0, Week 4, Week 12
  Schirmer test
Conjunctival staining | Day 0, Week 4, Week 12
  Oxford grading scale

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Kaercher, Dr., Principal Investigator — Praxis Dr. Thomas Kaercher
Locations (5):
- Germany (5):
  - Praxis Dr. Kaercher, Heidelberg, Baden-Wurttemberg
  - Praxis Prof. Dr. Anselm Kampik & Kollegen, Munich, Bavaria
  - Augenzentrum Olching, Olching, Bavaria
  - Augenheilkunde Lindenthal, Köln-Lindenthal, North Rhine-Westphalia
  - Dr. Flamm & Böker: Augenärzte am Tibarg, Hamburg

IPD SHARING:
Plan to Share IPD: No